CLINICAL TRIAL: NCT03905018
Title: Acute and Subacute Effect of Tadalafil Administration on Vasodilatation Mediated by Flow in Patients With Obesity Grade I-ii and Erectil Dysfunction
Brief Title: Effect of Tadalafil Administration on Vasodilatation Mediated by Flow in Patients With Obesity Grade I-II
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, Investigador principal, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDLF
Record Dates: First submitted 2019-02-19; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Obesity and Erectile Dysfuntion
MeSH Terms: conditions — Obesity | interventions — Tadalafil

STUDY DESIGN:
Intervention Model Description: A double-blind clinical trial with randomization and control group will be carried out. Male patients aged 25-60 years, BMI ≥30, without comorbidities will be included.
Who Masked: Participant, Investigator
Masking Description: A double-blind clinical trial with randomization and control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tadalafil (Experimental): Male patients aged 25-60 years, BMI ≥30, without comorbidities will be included. They should not be under treatment with iPDE5 or statins, nor should they have uncontrolled ischemic heart disease. To carry out this test, two groups will be created: the first will receive a single dose of tadalafil 20 mg orally
  Interventions: Drug: Tadalafil 20 MG
- calcined magnesia (placebo) (Placebo Comparator): Male patients aged 25-60 years, BMI ≥30, without comorbidities will be included. They should not be under treatment with iPDE5 or statins, nor should they have uncontrolled ischemic heart disease. To carry out this test, two groups will be created: the second will receive 20 mg of calcined magnesia (placebo),after a single administration
  Interventions: Drug: Tadalafil 20 MG

INTERVENTIONS:
Drug: Tadalafil 20 MG — tadalafil 20 mg orally ,after a single administration
  Other Names: tadalafil

SUMMARY:
Obesity is a public health problem, not only for its high prevalence, but also because of the comorbidities found in it. Within the physiopathological mechanisms associated with obesity is a low-grade inflammatory state that is associated with endothelial dysfunction Endothelial dysfunction is known to be the beginning of the atherosclerotic process that eventually leads to the development of cardiovascular disease.

Erectile dysfunction is an example of endothelial dysfunction, where blood flow is compromised as a consequence of a reduction in the production of nitric oxide among others.

Tadalafil, which is an inhibitor of PDE-5, is currently used as a treatment for erectile dysfunction. However, it has been observed that the administration of tadalafil in patients with éndothelial dysfunction decreases arterial stiffness, having a positive effect on it, in addition it reduces the pulse pressure, systolic and diastolic pressure.

DETAILED DESCRIPTION:
: The objective is to evaluate the effect of administration of tadalafil on vasodilatation mediated by flow in patients with obesity grade I-II and erectil dysfunction. A double-blind clinical trial with randomization and control group will be carried out. Male patients aged 25-60 years, BMI ≥30, without comorbidities will be included. They should not be under treatment with iPDE5 or statins, nor should they have uncontrolled ischemic heart disease. To carry out this test, two groups will be created: the first will receive a single dose of tadalafil 20 mg orally and the second will receive 20 mg of calcined magnesia (placebo),after a single administration, 24 hours later the investigators are going to evaluate vasodilatation mediated by. In addition, they will have a metabolic profile at the beginning.

For the analysis of results the statistical program SPSS version 21 for Windows will be used. The results will be expressed in averages and standard deviation and normality tests will be applied such as Kolmogorov Smirnof, Shapiro Wilk, as well as the Willcoxon and U Mann Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Age 25 to 60 years
* Obesity grade I-II
* .Sign the inform consent form.
* Answer the questionary IIFE

Exclusion Criteria:

. DM 1-2

* Systemic arterial hypertension
* Uncontrolled Mixed Dyslipidemia or under Hypolipemiant Treatment with statins.
* Active smoking
* Precedent of uncontrolled Ischemic cardiopathy.
* Use of anti-inflammatory drugs, including Acetylsalicylic acid, antihypertensive, antihyperglucemic, anti-anginal drugs, recent use of antiviral drugs that contains vasoconstrictors.
* Hepatic, renal, thyroid, and/or pulmonary decompensated disease.
* The precedent of hypersensibility to the phosphodiesterase-5 inhibitors.
* Patients that are under treatmen with iPDE

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male patients aged 25-60 years, BMI ≥30, without comorbidities will be included. They should not be under treatment with iPDE5 or statins, nor should they have uncontrolled ischemic heart disease
Enrollment: 80 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
vasodilatation mediated by flow | 24 hours
  the effect of administration of tadalafil on vasodilatation mediated by flow with UNEXEF in patients with obesity grade I-II and erectil dysfunction. A double-blind clinical trial with randomization and control group will be carried out.

SECONDARY OUTCOMES:
International Index Erectile Function | 24 hours
  evaluate erectile funtion with a test (IIFE)

CONTACTS AND LOCATIONS:
Locations (1):
- Fernando Grover Paez, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No